CLINICAL TRIAL: NCT02380690
Title: Evaluation of a Peer Coach-Led Intervention to Improve Pain Symptoms (ECLIPSE)
Brief Title: Evaluation of a Peer Coach-Led Intervention to Improve Pain Symptoms
Acronym: ECLIPSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 14-070; 1410626162 (Other: Indiana University)
Record Dates: First submitted 2015-02-23; First posted 2015-03-05 (Estimated); Results first posted 2020-08-17 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Chronic Pain
Keywords: self-management; peer support; social support
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peer Coach Assignment (Experimental): Veteran participants will be assigned to a peer coach, who delivered self-management instruction one-on-one over a 6-month period.
  Interventions: Behavioral: Peer Coach Assignment
- Control (No Intervention): Veteran participants will attend a 2-hour class in pain "basics" and pain self-management. Veterans will aso be given a set of pamphlets related to pain self-management.

INTERVENTIONS:
Behavioral: Peer Coach Assignment — Veterans will be assigned a peer coach to meet with for 6 months to discuss pain self-management.
  Arms: Peer Coach Assignment

SUMMARY:
To maximize implementation potential of pain self-management in the VA, alternative delivery methods are needed to provide Veterans with education and support needed to self-manage their pain, without requiring additional resources from healthcare teams. A novel and promising approach is a peer coaching model, in which Veterans with chronic pain who are successfully managing their pain offer information, support, and mentorship to other Veterans with pain.

DETAILED DESCRIPTION:
The investigators' goal is to test the effectiveness of a peer coaching model among Veterans. The investigators are examining feasibility for implementation alongside effectiveness, to shorten the timeline to implementation.

Aim 1 (primary aim): To compare 6-month (primary endpoint) and 9-month (sustained effects) effects of peer-supported chronic pain self-management versus controls on overall pain (intensity and function).

Hypothesis 1: Veterans in the peer support arm will experience reduced overall pain compared to controls.

Aim 2 (secondary aim): To compare 6- and 9-month effects of peer-supported chronic pain self-management versus controls on self-efficacy, social support, pain coping, patient activation, health-related quality of life, and health service utilization.

Hypothesis 2: Veterans in the peer support arm will experience greater self-efficacy, social support, pain coping, patient activation, and health-related quality of life, and lower health service utilization, compared to controls.

Aim 3 (pre-implementation aim): To explore facilitators and barriers to implementation of peer support for chronic pain, intervention costs, and fidelity to the model.

ELIGIBILITY:
Inclusion Criteria:

* have musculoskeletal pain in the low back, cervical spine, or extremities (hip, knee, or shoulder) for 3 months
* have at least moderate pain severity, defined by pain 5 on a 0 (no pain) to 10 (worst pain imaginable) scale
* indicate willingness to engage in phone or in-person contact on a regular basis with another Veteran

Exclusion Criteria:

* if the electronic medical record indicates a diagnosis of a psychotic disorder (e.g., International Classification of Diseases (ICD) ICD-9 codes 295-295.9 for schizophrenia)
* current substance dependence (e.g., ICD-9 codes 304-304.9)
* severe medical conditions precluding participation (e.g., New York Heart Association Class III or IV heart failure, ICD-9 codes 428-428.9 )
* if the eligibility screener given to prospective participants reveals active suicidal ideation severe hearing or speech impairment
* pending surgery for a musculoskeletal condition (e.g., back surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Sassi Matthias, PhD MS BA, Principal Investigator — Richard L. Roudebush VA Medical Center, Indianapolis, IN
Locations (1):
- Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon request, the Research Service will consider requests for the final data sets underlying the publications to be provided to the public. The limited dataset will include de-identified data relevant to the specific request. Independent research groups can view relevant data to evaluate the extent that data sources support conclusions made by authors in published studies as well as observe additional emergent themes and view supplemental details that might not be included in publications.
Supporting Information: Study Protocol, ICF
Time Frame: The data will become available once the study team completes all analyses.
Access Criteria: The Research Service will evaluate individual requests.

REFERENCES:
- [Result] Matthias MS, Daggy J, Adams J, Menen T, McCalley S, Kukla M, McGuire AB, Ofner S, Pierce E, Kempf C, Heisler M, Bair MJ. Evaluation of a peer coach-led intervention to improve pain symptoms (ECLIPSE): Rationale, study design, methods, and sample characteristics. Contemp Clin Trials. 2019 Jun;81:71-79. doi: 10.1016/j.cct.2019.04.002. Epub 2019 Apr 2. PMID 30951837
- [Result] Shue SA, McGuire AB, Matthias MS. Facilitators and Barriers to Implementation of a Peer Support Intervention for Patients with Chronic Pain: A Qualitative Study. Pain Med. 2019 Jul 1;20(7):1311-1320. doi: 10.1093/pm/pny229. PMID 30481295
- [Result] Matthias MS, Daggy J, Ofner S, McGuire AB, Kukla M, Bair MJ. Exploring peer coaches' outcomes: Findings from a clinical trial of patients with chronic pain. Patient Educ Couns. 2020 Jul;103(7):1366-1372. doi: 10.1016/j.pec.2020.02.007. Epub 2020 Feb 5. PMID 32044190
- [Result] Matthias MS, Bair MJ, Ofner S, Heisler M, Kukla M, McGuire AB, Adams J, Kempf C, Pierce E, Menen T, McCalley S, Johnson NL, Daggy J. Peer Support for Self-Management of Chronic Pain: the Evaluation of a Peer Coach-Led Intervention to Improve Pain Symptoms (ECLIPSE) Trial. J Gen Intern Med. 2020 Dec;35(12):3525-3533. doi: 10.1007/s11606-020-06007-6. Epub 2020 Jul 22. PMID 32700220
- [Derived] Matthias MS, Hirsh AT, Ofner S, Daggy J. Exploring the Relationships Among Social Support, Patient Activation, and Pain-Related Outcomes. Pain Med. 2022 Apr 8;23(4):676-685. doi: 10.1093/pm/pnab306. PMID 34718764

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants who enrolled withdrew prior to completing baseline assessments, leaving 119 randomized to the intervention and 94 to the control group.
Period: Overall Study
Arm/Group | Peer Coach Assignment | Control
Started | 119 | 94
Completed | 85 | 82
Not Completed | 34 | 12
Not completed — Lost to Follow-up | 14 | 4
Not completed — Withdrawal by Subject | 20 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peer Coach Assignment | Control | Total
Number analyzed (Participants) | 119 | 94 | 213
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (12.6) | 58.6 (13.3) | 56.8 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 16 | 40
  Male | 95 | 78 | 173
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 28 | 31 | 59
  White | 77 | 55 | 132
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 14 | 8 | 22
Region of Enrollment [Number; unit: participants]
  United States | 119 | 94 | 213
Brief Pain Inventory Total [Mean (Standard Deviation); unit: units on a scale] — Range: 0-10 (0 = no pain; 10 = worst pain imaginable)
  units on a scale | 5.8 (1.9) | 5.8 (1.9) | 5.8 (1.9)
Perceived Social Support [Mean (Standard Deviation); unit: units on a scale] — Range: 12-24 (higher numbers = greater social support)
  units on a scale | 62.2 (16.5) | 62.6 (18.1) | 62.3 (17.2)
Self-Efficacy [Mean (Standard Deviation); unit: units on a scale] — Range: 0-10 (higher numbers = higher self-efficacy)
  units on a scale | 6.1 (2.2) | 6.2 (2.3) | 6.1 (2.2)
Anxiety [Mean (Standard Deviation); unit: units on a scale] — Generalized Anxiety Disorder-7 (GAD-7, 0-21, higher numbers = higher anxiety)
  units on a scale | 6.1 (5.3) | 6.2 (5.4) | 6.1 (5.3)
Depression [Mean (Standard Deviation); unit: units on a scale] — Patient Health Questionnaire (PHQ-8, 0-24, higher numbers = higher depression)
  units on a scale | 9.3 (6.4) | 8.9 (6.0) | 9.2 (6.2)
Pain Catastrophizing [Mean (Standard Deviation); unit: units on a scale] — Range: 0-52 (higher numbers = higher catastrophizing)
  units on a scale | 20.8 (13.1) | 21.5 (13.3) | 21.1 (13.2)
Patient Activation [Mean (Standard Deviation); unit: units on a scale] — Patient Activation Measure (0-100, higher numbers = higher activation)
  units on a scale | 60.6 (13.5) | 57.9 (13.8) | 59.4 (13.7)
General Health Perceptions [Mean (Standard Deviation); unit: units on a scale] — SF-36 (Range: 0-100, higher numbers equal higher health perceptions)
  units on a scale | 52.2 (20.9) | 52.8 (21.1) | 52.5 (21.0)

OUTCOME MEASURES:

1. Primary Outcome: Brief Pain Inventory (BPI) (Overall Pain Assessment)
Description: The BPI was developed to assess the severity of pain and the impact of pain on daily functioning, and has been validated in primary care studies. (Range = 0-10, 0 = no pain, 10 = worst pain imaginable)
Time Frame: 6 months
Population: 21 withdrew and 14 were lost to follow up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Coach Assignment | Control
Number analyzed (Participants) | 92 | 86
units on a scale | 5.6 (2.0) | 5.6 (1.9)
Statistical Analysis 1: Comparison: Peer Coach Assignment vs Control; Test type: Superiority — ECLIPSE was powered to detect an effect size of 0.45; p = 0.981, Regression, Linear — Statistical significance was set at p<0.05

2. Primary Outcome: Brief Pain Inventory (BPI) (Overall Pain Assessment)
Description: as for outcome 1
Time Frame: 9 months
Population: 7 withdrew and 4 were lost to follow up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Coach Assignment | Control
Number analyzed (Participants) | 85 | 82
units on a scale | 5.4 (2.0) | 5.3 (2.0)
Statistical Analysis 1: Comparison: Peer Coach Assignment vs Control; Test type: Superiority; p = 0.774, Regression, Linear

3. Secondary Outcome: Pain Catastrophizing
Description: Pain Catastrophizing Scale, a 13-item scale that assesses catastrophizing - a pain belief that has been found to be a strong predictor of poor treatment response. (Range: 0-52, higher numbers = higher catastrophizing)
Time Frame: 6 months
Population: 21 withdrew and 14 lost to follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Coach Assignment | Control
Number analyzed (Participants) | 92 | 86
units on a scale | 21.8 (13.8) | 22.0 (11.8)
Statistical Analysis 1: Comparison: Peer Coach Assignment vs Control; Test type: Superiority — Power was based on primary outcome; p = 0.999, Regression, Linear — Statistical significance was set at p<0.05. A Sidak adjustment was used to account for multiple comparisons. Unadjusted p-value = 0.546

4. Secondary Outcome: Perceived Social Support
Description: Measures perceptions of social support.(Range: 12-84, higher numbers = higher perceptions of social support)
Time Frame: 6 months
Population: 21 withdrew and 14 lost to follow up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Coach Assignment | Control
Number analyzed (Participants) | 92 | 86
units on a scale | 62.0 (17.9) | 60.4 (16.4)
Statistical Analysis 1: Comparison: Peer Coach Assignment vs Control; Test type: Superiority; p = 0.999, Regression, Linear — Statistical significance was set at p<0.05. A Sidak adjustment was used to account for multiple comparisons. Unadjusted p-value = 0.403

5. Secondary Outcome: Perceived Social Support
Description: Measures perceptions of social support.(Range: 12-84, higher numbers = higher perceptions of social support)
Time Frame: 9 months
Population: 7 withdrew and 4 were lost to follow up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Coach Assignment | Control
Number analyzed (Participants) | 85 | 82
units on a scale | 63.6 (17.8) | 62.1 (17.3)
Statistical Analysis 1: Comparison: Peer Coach Assignment vs Control; Test type: Superiority; p = 0.999, Regression, Linear — Statistical significance was set at p<0.05. A Sidak adjustment was used to account for multiple comparisons. Unadjusted p-value = 0.452

6. Secondary Outcome: Self Efficacy
Description: Adapted from the Arthritis Self Efficacy Scale (Range 0-10, higher numbers = higher self efficacy)
Time Frame: 6 months
Population: 21 withdrew and 14 lost to follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Coach Assignment | Control
Number analyzed (Participants) | 92 | 86
units on a scale | 6.3 (2.3) | 6.1 (2.1)
Statistical Analysis 1: Comparison: Peer Coach Assignment vs Control; Test type: Superiority; p = 0.980, Regression, Linear — Statistical significance was set at p<0.05. A Sidak adjustment was used to account for multiple comparisons. Unadjusted p-value = 0.243

7. Secondary Outcome: Self Efficacy
Description: Adapted from the Arthritis Self Efficacy Scale (Range 0-10, higher numbers = higher self efficacy)
Time Frame: 9 months
Population: 7 withdrew and 4 lost to follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Coach Assignment | Control
Number analyzed (Participants) | 85 | 82
units on a scale | 6.4 (2.2) | 6.1 (2.2)
Statistical Analysis 1: Comparison: Peer Coach Assignment vs Control; Test type: Superiority; p = 0.864, Regression, Linear — Statistical significance was set at p<0.05. A Sidak adjustment was used to account for multiple comparisons. Unadjusted p-value = 0.133

8. Secondary Outcome: Anxiety
Description: GAD-7 (Range 0-21, higher numbers = higher anxiety)
Time Frame: 6 months
Population: 21 withdrew and 14 lost to follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Coach Assignment | Control
Number analyzed (Participants) | 92 | 86
units on a scale | 6.9 (5.4) | 6.2 (4.9)
Statistical Analysis 1: Comparison: Peer Coach Assignment vs Control; Test type: Superiority; p = 0.780, Regression, Linear — Statistical significance was set at p<0.05. A Sidak adjustment was used to account for multiple comparisons. Unadjusted p-value = 0.102

9. Secondary Outcome: Anxiety
Description: GAD-7 (Range 0-21, higher numbers = higher anxiety)
Time Frame: 9 months
Population: 7 withdrew and 4 lost to follow up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Coach Assignment | Control
Number analyzed (Participants) | 85 | 82
units on a scale | 6.5 (5.5) | 6.4 (5.3)
Statistical Analysis 1: Comparison: Peer Coach Assignment vs Control; Test type: Superiority; p = 0.999, Regression, Linear — Statistical significance was set at p<0.05. A Sidak adjustment was used to account for multiple comparisons. Unadjusted p-value = 0.536

10. Secondary Outcome: Depression
Description: PHQ-8 (Range: 0-24, higher numbers = higher depression)
Time Frame: 6 months
Population: 21 withdrew and 14 lost to follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Coach Assignment | Control
Number analyzed (Participants) | 92 | 86
units on a scale | 10.1 (6.7) | 9.1 (5.4)
Statistical Analysis 1: Comparison: Peer Coach Assignment vs Control; Test type: Superiority; p = 0.997, Regression, Linear — Statistical significance was set at p<0.05. A Sidak adjustment was used to account for multiple comparisons. Unadjusted p-value = 0.340

11. Secondary Outcome: Depression
Description: PHQ-8 (Range: 0-24, higher numbers = higher depression)
Time Frame: 9 months
Population: 7 withdrew and 4 lost to follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Coach Assignment | Control
Number analyzed (Participants) | 85 | 82
units on a scale | 9.2 (6.2) | 8.3 (5.8)
Statistical Analysis 1: Comparison: Peer Coach Assignment vs Control; Test type: Superiority; p = 0.999, Regression, Linear — Statistical significance was set at p<0.05. A Sidak adjustment was used to account for multiple comparisons. Unadjusted p-value = 0.384

12. Secondary Outcome: Pain Catastrophizing
Description: as for outcome 3
Time Frame: 9 months
Population: 7 withdrew and 4 lost to follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Coach Assignment | Control
Number analyzed (Participants) | 85 | 82
units on a scale | 19.0 (13.5) | 20.5 (12.4)
Statistical Analysis 1: Comparison: Peer Coach Assignment vs Control; Test type: Superiority; p = 0.999, Regression, Linear — Statistical significance was set at p<0.05. A Sidak adjustment was used to account for multiple comparisons. Unadjusted p-value = 0.730

13. Secondary Outcome: Patient Activation
Description: Patient Activation Measure (Range: 0-100, higher numbers = higher activation)
Time Frame: 6 months
Population: 21 withdrew and 14 lost to follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Coach Assignment | Control
Number analyzed (Participants) | 92 | 86
units on a scale | 63.5 (14.9) | 58.7 (14.3)
Statistical Analysis 1: Comparison: Peer Coach Assignment vs Control; Test type: Superiority; p = 0.914, Regression, Linear — Statistical significance was set at p<0.05. A Sidak adjustment was used to account for multiple comparisons. Unadjusted p-value = 0.161

14. Secondary Outcome: Patient Activation
Description: Patient Activation Measure (Range: 0-100, higher numbers = higher activation)
Time Frame: 9 months
Population: 7 withdrew and 4 were lost to follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Coach Assignment | Control
Number analyzed (Participants) | 85 | 82
units on a scale | 62.8 (14.7) | 60.5 (14.9)
Statistical Analysis 1: Comparison: Peer Coach Assignment vs Control; Test type: Superiority; p = 0.999, Regression, Linear — Statistical significance was set at p<0.05. A Sidak adjustment was used to account for multiple comparisons. Unadjusted p-value = 0.930

15. Secondary Outcome: General Health Perceptions
Description: SF-36 General Health Perceptions (Range: 0-100, higher numbers = higher health perceptions)
Time Frame: 6 months
Population: 21 withdrew and 14 lost to follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Coach Assignment | Control
Number analyzed (Participants) | 92 | 86
units on a scale | 52.7 (21.7) | 50.1 (19.7)
Statistical Analysis 1: Comparison: Peer Coach Assignment vs Control; Test type: Superiority; p = 0.999, Regression, Linear — Statistical significance was set at p<0.05. A Sidak adjustment was used to account for multiple comparisons. Unadjusted p-value = 0.379

16. Secondary Outcome: General Health Perceptions
Description: SF-36 General Health Perceptions (Range: 0-100, higher numbers = higher health perceptions)
Time Frame: 9 months
Population: 7 withdrew and 4 were lost to follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Coach Assignment | Control
Number analyzed (Participants) | 85 | 82
units on a scale | 50.9 (21.5) | 51.9 (21.0)
Statistical Analysis 1: Comparison: Peer Coach Assignment vs Control; Test type: Superiority; p = 0.999, Regression, Linear — Statistical significance was set at p<0.05. A Sidak adjustment was used to account for multiple comparisons. Unadjusted p-value = 0.969

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Peer Coach Assignment | Control
All-Cause Mortality (participants affected / at risk) | 0/119 | 0/94
Serious Adverse Events (participants affected / at risk) | 0/119 | 0/94
Other Adverse Events (participants affected / at risk) | 0/119 | 0/94

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT02380690/Prot_SAP_000.pdf